CLINICAL TRIAL: NCT02288689
Title: Clinical and Sonoelasographic Evaluation of the Elasticity of the Uterine Cervix in Pregnant Patients at Term
Acronym: EUC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Rami Aviram, MD, Meir Medical Center
Other Study IDs: 0180-14-MMC
Record Dates: First submitted 2014-10-26; First posted 2014-11-11 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Acuuvix SonoAce UGEO — Ultrasonographic vaginal examination

SUMMARY:
In this study the investigators aim to compare the cervical dilation time in pregnant patients at term who had clinical evaluation of the cervical consistency with patients who had also quantitative measurement of the cervical elasticity in .

DETAILED DESCRIPTION:
Softening of the uterine cervix in pregnant patients at term is usually evaluated clinically by subjective vaginal manual examination (Bishop's score).One of the variables of the score is cervical consistency which is considered important factor.The cervical consistency is described as soft,medium or stiff.However, the digital assessment of consistency is subjective and less reproducible.The Bishop's score also gives information about expected duration of labor after induction. The consistency of the uterine cervix can also be evaluated objectively sonoelastographically by measuring the cervical elasticity.This is illustrated by a color map, where low stiffness (soft tissue) is indicated in red, middle stiffness is in green and high stiffness (hard tissue) is in blue.In this study we aim to compare the cervical dilation time between the clinical evaluation of the cervical consistency and the quantitative measurement of the cervical elasticity in pregnant patients at term.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients at term

Exclusion Criteria:

* Various pregnancy complications

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients 20-44 years old at term
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Assess elasticity of uterine cervix through comparison of sonoelastographic evaluation and manual vaginal examination [Bishop Score] in pregnant patients at term | at time of the manual vaginal examination and participants will be followed for the duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rami Aviram, MD, Principal Investigator — Meir Medical Center